CLINICAL TRIAL: NCT02632812
Title: Double-blind Trial on the Gastrointestinal Integrity Evaluation After Daily Naproxen 1100 mg + Rebamipide 200mg for 7 Days Versus Naproxen 1100mg + Placebo for 7 Days
Brief Title: Gastrointestinal Integrity After Naproxen + Rebamipide Versus Naproxen + Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 025/14
Record Dates: First submitted 2015-11-23; First posted 2015-12-17 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Gastrointestinal Lesions
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebamipide & Naproxen (Experimental): Rebamipide 100 mg effervescent granules (oral) Twice daily (total dose = 200 mg) for 7 days
  Interventions: Drug: Rebamipide effervescent granules; Drug: Naproxen tablet
- Placebo & Naproxen (Placebo Comparator): Sugar pill manufactured to mimic Rebamipide 100 mg effervescent granules (oral) Twice daily for 7 days
  Interventions: Drug: Placebo effervescent granules; Drug: Naproxen tablet

INTERVENTIONS:
Drug: Rebamipide effervescent granules — Rebamipide effervescent granules 100mg (oral), twice daily for 7 days
  Arms: Rebamipide & Naproxen
Drug: Placebo effervescent granules — Placebo effervescent granules (oral), twice daily for 7 days
  Arms: Placebo & Naproxen
Drug: Naproxen tablet — Naproxen tablet 550mg (tablet), twice daily for 7 days

SUMMARY:
This is a double-blind, placebo-controlled, randomized, parallel trial to evaluate if rebamipide reduces the number of gastric events caused by naproxen. Sample size is 24 participants (12 per treatment group), male or female, aged 18 years-old and above.

Primary objective is to compare rebamipide effervescent granules 100 mg twice daily, plus naproxen (coated tablets) 550 mg twice daily to placebo plus naproxen 550 mg twice daily, for seven days, in reduction of gastric events caused by naproxen. Secondary objective is to evaluate safety and tolerability of rebamipide after multiple administrations.

Participants will receive either rebamipide + naproxen or placebo + naproxen, as above, during 7 consecutive days, which will be accompanied by a follow-up visit.

Gastric integrity will be assessed, before and after treatment, by endoscopy, with stomach biopsies and detection of H. pylori. Additionally, detection of occult blood in the stool will be performed, before and after treatment.

From the above-mentioned biopsies, dosage of prostaglandin E2 and histopathological analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female study participants, aged 18 years-old and above; women cannot be pregnant or breastfeeding;
* Body mass index (BMI) greater than or equal to 19 and less than or equal to 28.75 Kg/m2;
* Good health conditions or without significant diseases, according to best medical judgement, according to protocol requirements and study evaluations: medical history, blood pressure and heart rate measurements, physical examination, electrocardiogram (ECG) and screening laboratory tests;
* Ability to understand the nature and objectives of the trial, including risks and adverse events; willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Known hypersensitivity to the investigational products (naproxen or rebamipide) or chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug;
* Subject does not present intact superior gastrointestinal mucosa, i.e., presenting bleeding, ulcers and apparent injuries in baseline endoscopy;
* Subject has achlorhydria (intragastric pH > 6.5);
* History or presence of hepatic or gastrointestinal diseases, or other condition that interferes with drug absorption, distribution, excretion or metabolism;
* Chronic therapy with any drugs, except oral contraceptives;
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic or psychiatric disease; hypotension or hypertension, of any etiology, that requires pharmacological treatment; history of myocardial infarction, angina and/or heart failure;
* Occult blood in the stool before treatment;
* Electrocardiographic findings that, at investigator criteria, are not recommended for study participation;
* Deviations on screening laboratory results that are considered as clinically relevant by the principal investigator;
* History of drugs and alcohol addiction or excessive alcohol consumption (> 35 g/day);
* Use of regular medications within 2 weeks prior study enrollment or use of any medications within one week prior to study enrollment, except oral contraceptives or cases which, based on drug's or metabolite's half-life, complete elimination can be assumed;
* Treatment, within 6 months before the trial, with any drugs known to have a well-established toxic potential to major organs;
* Participation in any other experimental research or administration of any experimental drug within 6 months before this trial;
* Any condition, according to investigator's best judgement, that prevents the subject to participate in the trial;
* Pregnancy, labor or miscarriage with 12 weeks before admission predicted date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Ltda.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gagliano-Juca T, Moreno RA, Zaminelli T, Napolitano M, Magalhaes AF, Carvalhaes A, Trevisan MS, Wallace JL, De Nucci G. Rebamipide does not protect against naproxen-induced gastric damage: a randomized double-blind controlled trial. BMC Gastroenterol. 2016 Jun 4;16(1):58. doi: 10.1186/s12876-016-0472-x. PMID 27259970

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebamipide 200 mg: Rebamipide 100 mg effervescent granules (oral) Twice daily (total dose = 200 mg)
  Rebamipide effervescent granules
  Naproxen tablet
- Placebo: Placebo effervescent granules (oral) Twice daily
  Placebo effervescent granules
  Naproxen tablet
Period: Overall Study
Arm/Group | Rebamipide 200 mg | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebamipide 200 mg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23.5 [18 to 49] | 28.5 [19 to 49] | 24.5 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Score - Cryer Score
Description: Cryer score according to gastroduodenal mucosal injury:
  0 = Normal or erythema
  1. = Any amount of submucosal hemorrhage or edema without erosions
  2. = 1 erosion +- submucosal hemorrhage or edema
  3. = 2-4 erosions +- submucosal hemorrhage or edema
  4. = 5 or more erosions and/or a single ulcer +- submucosal hemorrhage or edema
  5. = Multiple ulcers +- submucosal hemorrhage or edema - Ulcer
Time Frame: 8 days
Population: All recruited volunteers completed the trial.
Measure: Median (Full Range); unit: Cryer score
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
Cryer score | 4 [0 to 5] | 4 [0 to 5]

2. Primary Outcome: Endoscopic Score - Modified Lanza Score
Description: Modified Lanza score according to gastroduodenal mucosal injury:
  0 = No hemorrhage or erosion observed
  1. = One or two hemorrhages or erosions observed in one gastric area
  2. = Three to five hemorrhages or erosions observed in one gastric area
  3. = Hemorrhages or erosions observed in two gastric areas, six or more hemorrhages or erosions observed in one gastric area, with the total number not exceeding ten in the entire stomach
  4. = Hemorrhages or erosions observed in three or more gastric areas; eleven or more hemorrhages or erosions observed widely in the entire stomach
  5. = Ulcer
Time Frame: 8 days
Measure: Median (Full Range); unit: Modified Lanza score
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
Modified Lanza score | 3.5 [0 to 5] | 4 [0 to 5]

3. Primary Outcome: Histopathological Score
Description: Histopathologic grade score developed for microscopic injury evaluation 0 = Normal gastric mucosa or mild chronic inflammation
  1. = Chronic gastritis without activity
  2. = Chronic gastritis with activity on antrum
  3. = Chronic gastritis with activity on the body
  4. = Chronic gastritis with activity on antrum and on the body
Time Frame: 8 days
Measure: Median (Full Range); unit: Histopathologic grade score
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
Histopathologic grade score
  Basal endoscopy | 1 [0 to 4] | 1 [0 to 4]
  End of treatment endoscopy | 1 [0 to 4] | 1 [0 to 4]

4. Primary Outcome: Intragastric pH
Time Frame: 8 days
Population: Intragastric PH measurement was not performed and for this reason it will not be available.
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Presence of H. Pylori by Biopsy
Description: Giemsa stain was used to diagnose H. pylori (positive = presence of H. pylori)
Time Frame: 8 days
Measure: Number; unit: participants
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
participants
  Basal endoscopy | 5 | 5
  End of treatment endoscopy | 6 | 6

6. Primary Outcome: Prostaglandin Level (PGE2 Quantification)
Description: Tissue prostaglandin concentration quantified by enzyme-linked immunosorbent assay (ELISA) using Cayman Chemical Monoclonal Prostaglandin E2 EIA Kit (item number 514010)
Time Frame: 8 days
Measure: Mean (95% Confidence Interval); unit: pg/mL (mean tissue PGE2 concentration)
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
pg/mL (mean tissue PGE2 concentration)
  Basal PGE2 concentration | 999 [890 to 1108] | 1005 [876 to 1134]
  End of treatment PGE2 concentration | 168 [155 to 181] | 241 [200 to 282]

7. Secondary Outcome: Number of Adverse Events
Time Frame: 60 days
Measure: Number; unit: adverse events
Arm/Group | Rebamipide & Naproxen | Placebo & Naproxen
Number analyzed (Participants) | 12 | 12
adverse events | 7 | 7

ADVERSE EVENTS:
Arm/Group | Rebamipide 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebamipide 200 mg (N=12) | Placebo (N=12)
Addominal distress (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Heartburn (Gastrointestinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No